CLINICAL TRIAL: NCT06323564
Title: Exploring How Emotional Intelligence and Cognitive Flexibility Affect the Measurement of Emotional Valence and Arousal in Two Populations: Patients With Anorexia Nervosa and Parkinson's Disease.
Brief Title: Exploring Emotional Intelligence and Cognitive Flexibility in Anorexia Nervosa and Parkinson's Disease.
Acronym: INTELLEGO
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 21C223
Record Dates: First submitted 2024-03-04; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Anorexia Nervosa; Parkinson Disease
Keywords: Emotional intelligence; Cognition; Emotional valence; Anorexia nervosa; Parkinson's disease
MeSH Terms: conditions — Anorexia Nervosa; Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson Disease (PD): The trial will be divided into two periods T0 (first evaluation at the time of admission to hospital) and T1 (15 days after T0, during rehabilitation period in hospital for patients with Parkinson's disease).
  First, as soon as patients are admitted to acute care,neuropsychological tests and self-report questionnaires will be administered.
  Subsequently, at both T0 and T1, standardized emotional images from the International Affective Picture System (IAPS) will be administered. For the entire duration of the test, peripheral physiological parameters such as ECG, BVP, GSR, EOG, RSP and facial EMG (corrugator and zygomaticus) will also be detected, as objective measures of emotional arousal (T0-T1).
  Interventions: Diagnostic Test: Neuropsychological tests in PD; Diagnostic Test: Self-report questionnaires in PD; Device: International Affective Picture System (IAPS)
- Anorexia Nervosa (AN): The trial will be divided into two periods T0 (first evaluation at the time of admission to hospital) and T1 (4 weeks after T0, during rehabilitation period in hospital.
  First, as soon as patients are admitted to acute care, neuropsychological tests and self-report questionnaires will be administered.
  Subsequently, at both T0 and T1, standardized emotional images from the International Affective Picture System (IAPS) will be administered. For the entire duration of the test, peripheral physiological parameters such as ECG, BVP, GSR, EOG, RSP and facial EMG (corrugator and zygomaticus) will also be detected, as objective measures of emotional arousal (T0-T1). Furthermore, the analysis of bio-humoral parameters (interleukin 6, cortisol, serotonin, catecholamines and endorphins) will be also performed through morning venous blood sampling at T0, at half of the rehabilitation process and at T1.
  Interventions: Device: International Affective Picture System (IAPS); Diagnostic Test: Neuropsychological tests in AN; Diagnostic Test: Self-report questionnaires in AN; Diagnostic Test: Analysis of bio-humoral parameters

INTERVENTIONS:
Diagnostic Test: Neuropsychological tests in PD — Colored Progressive Matrices (BDM), Stroop Test (Caffarra et al., 2000), Stroop Test (Caffarra et al., 2000), Attentional Matrices (part I - Della Sala et al., 1992), Attentional Matrices (part The - Della Sala et al., 1992), Trail Making Test (Giovagnoli et al., 1996 - part A), Trail Making Test (Giovagnoli et al., 1996 - part B), Trail Making Test (Giovagnoli et al., 1996 - B-A), MMSE (Grigoletto et al., 1999), Clock Drawing - PD (Caffarra et al., 2011), Digit Span Forward (Orsini et al., 1987), Digit Span Backward (Monaco et al. , 2012), 15 Rey Words - Immediate Recall (BDM), 15 Rey Words - Deferred Recall (BDM), Phonemic Fluency (Costa et al., 2014), Semantic Fluency (Costa et al., 2014), Frontal Assessment Battery ( FAB - Apollonio et al.,2005).
  Groups: Parkinson Disease (PD)
Diagnostic Test: Self-report questionnaires in PD — STAI Y2 (trait anxiety), TEIque (153 items), STAI Y1 (state anxiety), ERQ (10 items), EISR (33 items), BDI (21 items), WLEIS (16 ITEMS), CFI (20 ITEMS ), CCFQ (18 ITEM).
  Groups: Parkinson Disease (PD)
Device: International Affective Picture System (IAPS) — Subsequently, at both T0 and T1, standardized emotional images from the International Affective Picture System (IAPS) will be administered. The images will be chosen based on the arousal-valence parameters, eliminating those with stimuli that are too salient with respect to the disorders examined. The order of administration will be organized and randomized between subjects as follows: 24 blocks of 2 minutes and for each block there will be 12 images of 10 seconds each. For the entire duration of the test, peripheral physiological parameters such as ECG, BVP, GSR, EOG, RSP and facial EMG (corrugator and zygomaticus) will also be detected, as objective measures of emotional arousal (T0-T1).
Diagnostic Test: Neuropsychological tests in AN — Verbal Fluencies, Tower of London, TMT-A & B
  Groups: Anorexia Nervosa (AN)
Diagnostic Test: Self-report questionnaires in AN — STAI Y2 (20 items trait anxiety), TEIque (153 items), STAI Y1 (20 items state anxiety), DFlex (24 items), ERQ (10 items), EISR (33 items), BDI (21 items), TAS-20 (20 items), WLEIS (16 ITEMS), CFI (20 ITEMS), CCFQ (18 items).
  Groups: Anorexia Nervosa (AN)
Diagnostic Test: Analysis of bio-humoral parameters — the analysis of bio-humoral parameters (interleukin 6, cortisol, serotonin, catecholamines and endorphins) will be also performed through morning venous blood sampling at T0, at half of the rehabilitation process and at T1
  Groups: Anorexia Nervosa (AN)

SUMMARY:
The main aim of this study is to demonstrate how disorders characterized by different types of "inflexibility", cognitive-affective type for Anorexia nervosa and motor one for Parkinson's disease, have an impact on how emotional stimuli are processed and on the transition within emotional states.

DETAILED DESCRIPTION:
Although many psychometric models have been developed on emotions, affect measurements, which represent the measurement of behavioural, subjective and neuropsychophysiological changes associated with an emotional episode, still remains one of the most debated topics. Emotions are entities with blurred boundaries and with substantial idiosyncrasies that characterize their measurable manifestations. One of the most consolidated theoretical reference models for measuring affect is that of James Russel called the "Affective Core Model". According to this model, emotion arises when the undifferentiated and pre-reflective magma of affect (core affect) is attracted by an external (or internal) object that can be defined as emotigenic, i.e. capable of defining the nature of emotional experience by orienting it along two dimensions principal factors. The most used theoretical model for affect measurement is the one that describes an emotional episode in the light of two distinguishable continuous dimensions: that of hedonic value (identifies the degree of pleasantness of the emotional event), of a subjective nature, and that of arousal or psychophysiological activation. Although this model has been widely corroborated in various disciplines, there is still a lack of a clear description of the process that allows an individual to transition from one emotionally object-oriented state to another.

This project proposes and intends to validate a new modality of three-dimensional psychometric modeling of emotions, based on the intersection between the consolidated two-dimensional model of arousal-valence and a third purely cognitive component definable as mental flexibility, capable of including high-level cognitive processes, intrinsically connected with the emotional sphere, such as emotional intelligence (Emotional Intelligence, EI) and emotional regulation.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's Disease
* Anorexia nervosa
* Written informed consent

Exclusion Criteria:

* Other psychiatric disorders
* Acute infectious diseases
* Chronic inflammatory diseases
* Other Disorders of central nervous system
* Pregnancy or breastfeeding
* tachy or bradyarrhythmias, other cardiac rhythm alterations that compromise the study of heart rate variability

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by Parkinson's Disease and Anorexia Nervosa
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-01-13 (Actual); Primary Completion 2024-08-13 (Estimated); Study Completion 2025-01-13 (Estimated)

PRIMARY OUTCOMES:
Change in International Affective Picture System (IAPS) | At baseline T0 (hospital admission) and T1 (15 days after T0 for PD, 4 weeks after T0 for AN)
  Self-Assessment Manikin (SAM) scale. Range score for each image: 1-5 (IAPS test: 24 blocks of 2 minutes and for each block there will be 12 images of 10 seconds each).

SECONDARY OUTCOMES:
Change in self-report questionnaires - STAI | At baseline T0 (hospital admission) and T1 (15 days after T0 for PD, 4 weeks after T0 for AN)
  State-Trait Anxiety Inventory (STAI); score range 20-80
Change in self-report questionnaires - BDI | At baseline T0 (hospital admission) and T1 (15 days after T0 for PD, 4 weeks after T0 for AN)
  Beck's Depression Inventory (BDI); score range 0-63
Change in Heart rate variability | At baseline T0 (hospital admission) and T1 (15 days after T0 for PD, 4 weeks after T0 for AN)
  High frequency (range 0.15-0.40 hz)
  * Low frequency (range 00.4-0.15 hz)
  * Ratio Low frequency/High frequency
Change in analysis of bio-humoral parameters | At baseline T0 (hospital admission), after 2 weeks and T1 (4 weeks after T0 for AN)
  Serotonin in serum (range 30 - 200 ng/ml)

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Oggebbio, Italy